CLINICAL TRIAL: NCT01673815
Title: Video Diversion During Fundoscopic Exam in Children: A Randomized Controlled Trial
Brief Title: Video Diversion During Fundoscopic Exam in Children
Acronym: CAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H11-01885
Record Dates: First submitted 2012-08-20; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Other Disorders of Optic Disc, Bilateral
Keywords: optic disk; fundoscopy; pediatric; clinical examination
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1st: R eye video. 2nd: L eye no video (Experimental): The right eye will be examined first with video, followed by the left eye without video.
  Interventions: Other: Video (played on a computer monitor)
- 1st: R eye no video. 2nd: L eye video (Experimental): The right eye will be examined without video, followed by the left eye with video.
  Interventions: Other: Video (played on a computer monitor)
- 1st: L eye video. 2nd: R eye no video (Experimental): The left eye will be examined first with video, followed by the right eye without video.
  Interventions: Other: Video (played on a computer monitor)
- 1st: L eye no video. 2nd: R eye video (Experimental): The left eye will be examined first without video, followed by the right eye with video.
  Interventions: Other: Video (played on a computer monitor)

INTERVENTIONS:
Other: Video (played on a computer monitor) — The intervention is a video (of the patient or caregiver's choice) which is played on a computer monitor during the fundoscopic examination.

SUMMARY:
Fundoscopy is an important aspect of the neurological examination, but can be challenging in uncooperative children. This study explored whether viewing a video (selected by patient or caregiver) during eye examination improves the success, duration and ease of pediatric fundoscopy.

Hypothesis: Showing a short video clip during a fundoscopic exam will increase the probability of successfully visualizing the optic disk and reduce the amount of time needed to perform a fundoscopic exam in children between 1-8 years old.

DETAILED DESCRIPTION:
The purpose of this study is to examine whether showing a video clip with sound of the patient's choice can improve the ease of fundoscopic exam as defined by improved success of visualizing the optic disk and the reduction in time needed to perform the exam. The investigators will also examine the physician's and caregiver's perception on whether the video was effective in improving the ease of the exam. The purpose of the video is to capture the visual attention of the patient thereby allowing the physician to swiftly perform the fundoscopic exam. The literature has suggested that young patients are most uncooperative, therefore the investigators will focus our study on younger patients 1-8 years old.

ELIGIBILITY:
Inclusion Criteria:

* 1-8 years old
* Capable of visualizing the video monitor
* Patient has 2 examinable eyes

Exclusion Criteria:

* Blind patient
* Patients < 1 or > 8 years old

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Success rate of visualizing the optic disk within 60 seconds | At the time of fundoscopy exam
  To determine whether showing a video clip with sound of the patient's choice can improve the success of fundoscopic exam in children as defined by the ability to visualize the optic disk within 60 seconds.

SECONDARY OUTCOMES:
Reduction in the amount of time needed to visualize the optic disk. | At the time of fundoscopy exam
  To determine whether showing a video clip with sound of the patient's choice can reduce the amount of time needed to perform a successful fundoscopic exam.
Improvement in the physician's and caregiver's (parent/legal guardian) perception of the ease of the fundoscopic exam. | At the time of fundoscopy exam
  Improvement in the physician's and caregiver's (parent/legal guardian) perception of the ease of the fundoscopic exam as determined by a 10 point likert scale (1 being easiest and 10 being hardest).

CONTACTS AND LOCATIONS:
Overall Officials: Ash Singhal, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Jan MM. Neurological examination of difficult and poorly cooperative children. J Child Neurol. 2007 Oct;22(10):1209-13. doi: 10.1177/0883073807306262. PMID 17940248
- [Background] Cok OY. Anaesthesia for eye examination. Current Anaesthesia & Critical Care 2008 February 2009;20(1):46.
- [Background] de la Barra F, Toledo V, Rodriguez J. Prediction of behavioral problems in Chilean schoolchildren. Child Psychiatry Hum Dev. 2005 Spring;35(3):227-43. doi: 10.1007/s10578-004-6459-9. PMID 15731888
- [Background] Colares V, Richman L. Factors associated with uncooperative behavior by Brazilian preschool children in the dental office. ASDC J Dent Child. 2002 Jan-Apr;69(1):87-91, 13. PMID 12119822
- [Background] Hussein MA, Coats DK, Paysse EA. Use of the RetCam 120 for fundus evaluation in uncooperative children. Am J Ophthalmol. 2004 Feb;137(2):354-5. doi: 10.1016/S0002-9394(03)00867-5. PMID 14962432